CLINICAL TRIAL: NCT01550081
Title: Exercise Intensity and Target Heart Rate During Aerobic Interval Training in Cardiac Rehabilitation
Brief Title: Target Heart Rate and Aerobic Interval Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: 2011/2632
Record Dates: First submitted 2012-03-07; First posted 2012-03-09 (Estimated); Last update posted 2013-11-28 (Estimated); Status verified 2013-11

CONDITIONS: Coronary Artery Disease
Keywords: exercise intensity; aerobic interval training; cardiac rehabilitation; group exercise
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rate of perceived exertion (Active Comparator): Exercise intensity controlled by Borg
  Interventions: Other: Rate of perceived exertion; Other: Heart rate monitor
- Heart rate monitor (Active Comparator): Exercise intensity controlled by heart rate monitors
  Interventions: Other: Heart rate monitor

INTERVENTIONS:
Other: Rate of perceived exertion — Exercise intensity controlled by Borg scale
  Arms: Rate of perceived exertion
Other: Heart rate monitor — Exercise intensity controlled by heart rate monitors

SUMMARY:
Aerobic interval training is shown to be superior in increasing oxygen uptake in both healthy and patients with coronary artery disease (CAD), compared to moderate continuous training. However, in cardiac rehabilitation exercise groups, exercise intensity is usually controlled with perceived exertion (Borg scale). The investigators will investigate degree of agreement between target heart rate and perceived exertion during interval training in cardiac rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* referred to cardiac rehabilitation
* able to perform exercise treadmill test

Exclusion Criteria:

* unstable angina
* severe arrhythmias
* heart failure

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2012-03; Primary Completion 2012-08 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
degree of agreement between target heart rate (THR) and perceived exertion | up to 1 hour
  Exercise intensity during one-hour exercise session monitored by Borg, subsequently one-hour exercise session monitored by heart rate monitor

CONTACTS AND LOCATIONS:
Overall Officials: Inger-Lise Aamot, MSc, Principal Investigator — Norwegian University of Science and Technology
Locations (1):
- Department of circulation and medical imaging, NTNU, Trondheim, Sør-Trøndelag, Norway

REFERENCES:
- [Result] Aamot IL, Forbord SH, Karlsen T, Stoylen A. Does rating of perceived exertion result in target exercise intensity during interval training in cardiac rehabilitation? A study of the Borg scale versus a heart rate monitor. J Sci Med Sport. 2014 Sep;17(5):541-5. doi: 10.1016/j.jsams.2013.07.019. Epub 2013 Aug 8. PMID 23988787